CLINICAL TRIAL: NCT02733705
Title: A Randomised Controlled Trial Comparing Combined Intravenous Propofol and Fentanyl Versus Intravenous Propofol Alone for Sedation in Patients Undergoing Transrectal Ultrasound-guided (TRUS) Prostate Biopsy
Brief Title: Intravenous Propofol and Fentanyl vs Propofol for Sedation in TRUS Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRUS
Record Dates: First submitted 2016-03-27; First posted 2016-04-11 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pain
Keywords: Pain; TRUS biopsy
MeSH Terms: conditions — Pain | interventions — Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): normal saline IV plus propofol infusion
  Interventions: Other: Control; Drug: propofol
- Fentanyl (Active Comparator): 0.5 mcg/kg ideal body weight IV plus propofol infusion
  Interventions: Drug: Fentanyl; Drug: propofol

INTERVENTIONS:
Other: Control — normal saline IV
  Arms: Control
Drug: Fentanyl — fentanyl 0.5 mcg/kg ideal BW
  Arms: Fentanyl
Drug: propofol — propofol infusion

SUMMARY:
Nowadays, TRUS biopsy become one of the most popular tests for diagnosis of prostate cancer. This procedure causes pain to the patients who does not received the sedative drugs or analgesic drugs. There are many ways to reduce pain and inconvenience for the patients, such as intravenous propofol, intravenous fentanyl etc. In Siriraj hospital, anesthesiologists usually give intravenous propofol with intravenous opioids but the visual analogue score after this procedure was average at 0.9-2.9. Furthermore, some systematic reviews have shown that there was no difference in pain score between periprostatic nerve block plus opioid and periprostatic nerve block only. So, this study is to find out whether opioids is need for TRUS biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 year
* Patient American society of anesthesiology physical status I-III.
* Scheduled for Transrectal ultrasound-guided prostate biopsy
* BMI equal to or less than 30 kg/cm2

Exclusion Criteria:

* Known hypersensitivity to propofol or fentanyl
* History of bleeding tendency
* Known case of active anal or rectal disease
* Unable to rate pain score
* History of drug abuse
* Chronic opioid use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Pain assess using Numeric rating scale (NRS) score | 20 minutes

SECONDARY OUTCOMES:
Number of participants with hypoxia defined as oxygen saturation <92% | 60 minutes
  The investigators define hypoxia as oxygen saturation < 92%. The investigators will report as number of episode.
Number of participants with hypotension, defined as systolic blood pressure <90 mmHg | 60 minutes
  The investigators define hypotension as systolic blood pressure< 90 mmHg. The investigators will report as number of episode.

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, Principal Investigator — Mahidol University
Locations (1):
- Sirilak Suksompong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suksompong S, Limratana P, Saengsomsuan N, Wongsawang N, Chaikittisilpa N. Propofol with or without fentanyl for pain relief after transrectal ultrasound-guided prostate (TRUS-P) biopsy: a randomized controlled study. Braz J Anesthesiol. 2021 Jul-Aug;71(4):345-351. doi: 10.1016/j.bjane.2021.02.001. Epub 2021 Feb 3. PMID 34229860